CLINICAL TRIAL: NCT01766323
Title: Prospective Randomized Study Evaluating the Effects of Modafinil in Patients Receiving Oral Morphine for Pain Palliation
Brief Title: Palliative Morphine With or Without Concurrent Modafinil
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Rajendra Prasad Government Medical College (Other)
Responsible Party: Principal Investigator, Swaroop Revannasiddaiah, Principal Investigator, Dr. Rajendra Prasad Government Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ModMorphine
Record Dates: First submitted 2013-01-08; First posted 2013-01-11 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Cancer; Pain Palliation; Excessive Sleepiness
Keywords: Morphine; Palliation; Cancer; Hospice; Sleepiness; Modafinil
MeSH Terms: conditions — Neoplasms; Disorders of Excessive Somnolence; Sleepiness | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm Placebo (Placebo Comparator): Oral placebo b.i.d, along with the dose of oral morphine required for pain palliation
  Interventions: Drug: Placebo
- Arm-Modafinil (Active Comparator): Oral modafinil at a dose of 100mg b.i.d along with the dose of oral morphine required for pain palliation
  Interventions: Drug: Modafinil

INTERVENTIONS:
Drug: Modafinil — Oral modafinil at a dose of 100mg b.i.d along with the dose of oral morphine required for pain palliation
  Arms: Arm-Modafinil
Drug: Placebo — Oral placebo b.i.d, along with the dose of oral morphine required for pain palliation
  Arms: Arm Placebo

SUMMARY:
Oral morphine is often utilized as a convenient and effective method of achieving palliation of pain in the terminally ill cancer patients. However, at effective doses, a majority of patients do experience an undue amount of excessive sleepiness. Given the generally low expected survival periods among this patient population, the fact that morphine causes the patient to spend a significant period of remaining life in sleep, is often unacceptable for the patients and their families. Given the proven benefits of modafinil in conditions characterized by excessive sleepiness (such as with narcolepsy and shift-work disorder), the investigators designed a prospective placebo controlled randomized trial by the addition of modafinil at a dose of 200mg per day (in two divided doses) for eligible patients after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed and confirmed malignancy
* Able to orally consume tablets
* Blood Pressure: Systolic <144mmHg; Diastolic <92mmHg
* Normal blood sugar
* No active systemic infections
* Consenting
* Oral morphine being consumed as a part of terminal symptom palliation

Exclusion Criteria:

* Candidates receiving oral morphine for temporary pain management, such as being potential candidates for radical curative approaches in the future
* Poor performance status (Karnofsky Performance Status score <50)
* Prior history of hypertension, diabetes, tuberculosis, epilepsy
* Prior history of psychiatric and neurological illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-06 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Patient reported sleepiness scores | Three months from enrollment
  Patient reported sleepiness scores will be recorded as per a visual analogue scale with scores ranging from 1 (no unusual sleepiness) to 5 (unable to stay awake). Recordings will be done on the first day of intervention, and repeated recordings will be procured once every two weeks till a total of seven readings are obtained over a time span of 3 months.

SECONDARY OUTCOMES:
Mood changes | Three months from enrollment
  Patients will be requested to report their self-perceived mood status by choosing one of three discrete options (improvement, worsening, no change). Each patient will provide a total of three responses over a period of three months from enrollment (at the end of each month from enrollment).

CONTACTS AND LOCATIONS:
Overall Officials: Swaroop Revannasiddaiah, MD, Principal Investigator — Dr. Rajendra Prasad Government Medical College; Bangalore Institute of Oncology; Muninder K Negi, MD, Study Director — Dr. Rajendra Prasad Government Medical College; Indira Gandhi Medical College; Sridhar P Susheela, MD, Study Chair — Bangalore Institute of Oncology; Madhup Rastogi, MD, Study Chair — Ram Manohar Lohia Insitute of Medical Sciences; Manoj K Gupta, MD, Study Chair — Indira Gandhi Medical College, Shimla
Locations (1):
- Tanda Government Medical College and Hospital, Kangra, Himachal Pradesh, India